CLINICAL TRIAL: NCT02512757
Title: The AminoIndex™ Study - A Case-Control Study to Verify Diagnostic Performance of AminoIndex™ Technology
Brief Title: A Case-Control Study to Verify Diagnostic Performance of AminoIndex™ Technology
Status: Completed | Type: Observational
Sponsor: Innovis LLC (Industry)
Collaborators: Ajinomoto Co., Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Ajinomoto 2015-01
Record Dates: First submitted 2015-07-27; First posted 2015-07-31 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Lung Cancer
Keywords: Neoplasms, Lung; Pulmonary Neoplasms; Pulmonary Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects will consent to archiving and future analysis of their blood samples for up to twenty (20) years.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Patients with lung nodule(s) ≥ 6 mm but ≤ 35 mm that have been biopsied and diagnosed with primary lung cancer who have not yet initiated treatment of any kind for their lung cancer will contribute a fasting blood sample.
- Group 2: Patients whose most recent screening imaging is within 60 days who have lung nodule(s) ≥ 6 mm but ≤ 35 mm that have been biopsied and determined to not be cancerous OR that have demonstrated no nodule growth for >2 years by repeat CT imaging will contribute a fasting blood sample.
- Group 3: Patients who have undergone low-dose computed tomography (LDCT) or standard computed tomography (CT) or X-ray testing to screen for lung cancer with no nodules suspicious for lung cancer within 1 year prior to signing informed consent will contribute a fasting blood sample.

SUMMARY:
This is a prospective, multi-center study to evaluate the diagnostic performance characteristics of the AminoIndex™ technology among patients at high risk for developing lung cancer as compared with standard lung cancer screening and diagnostic procedures including low-dose CT, high-dose CT, biopsy and histopathology.

DETAILED DESCRIPTION:
This is a prospective, multi-center study to evaluate the diagnostic performance characteristics of the AminoIndex™ technology among patients at high risk for developing lung cancer as compared with standard lung cancer screening and diagnostic procedures including low-dose CT, high-dose CT, biopsy and histopathology.

The study will enroll patients into one of three arms:

1. patients with lung nodule(s) ≥ 6 mm but ≤ 35 mm that have been biopsied and diagnosed with primary lung cancer who have not yet initiated treatment of any kind for their lung cancer;
2. patients with lung nodule(s) ≥ 6 mm but ≤ 35 mm that have been biopsied and determined to not be cancerous OR that have demonstrated no nodule growth for > 2 years by repeat CT imaging; and
3. patients at high-risk for lung cancer (per NLST guidelines) with no evidence or history of lung cancer (negative LDCT/CT/X-ray).

ELIGIBILITY:
Inclusion Criteria

All Groups:

* Able to read, understand and sign informed consent to participate in study.
* Willing and able to provide written informed consent.
* Willing and able to meet all study requirements and undergo venipuncture to provide a fasting blood sample.

Group 1:

* Men or women age 18 years or older;
* Lung nodule size ≥ 6 mm but ≤ 35 mm/ lung, nodule or mass.
* Diagnosis of lung cancer based upon histopathology performed on lung nodule, lesion or mass tissue obtained from biopsy or surgical excision performed after study-related fasting blood sample obtained.

Group 2:

* Men or women age 18 years or older;
* Lung nodule size ≥ 6 mm but ≤ 35 mm/ lung nodule, lesion or mass;
* Definitive diagnosis of benign (non-cancerous) lung nodule based upon one of the following:

  * Histopathology performed on lung nodule tissue obtained from biopsy or surgical excision performed after study-related fasting blood sample obtained;
  * No nodule growth for > 2 years by repeat CT imaging, the most recent being performed within the 60 days prior to signing informed consent.

Group 3:

* Men or women age 55-79 years inclusive;
* Current smoker or quit < 15 years ago with a > 30 pack-year smoking history (equivalent of 1 pack per day for 30 or more years)*.
* Have undergone low-dose computed tomography (LDCT) or standard computed tomography (CT) or X-ray testing to screen for lung cancer with no nodules suspicious for lung cancer within 1 year prior to signing informed consent.

' * ' One pack year is calculated as follows: 20 cigarettes = 1 pack. One "pack year" is the equivalent of smoking:

* 20 cigarettes (one pack) per day for one year; or
* 40 cigarettes (two packs) per day for 6 months; or
* 60 cigarettes (three packs) per day for 3 months

Exclusion Criteria

* Inability to fast for 8 hours prior to the blood sample collection.
* Known to be positive for HIV and/or, HBV and/or HCV.
* Pregnancy.
* Breastfeeding.
* Currently undergoing dialysis.
* Congenital metabolic disease.
* Currently receiving investigational treatments of any type.
* History of receiving any drug therapy or surgery for the treatment of lung cancer.
* Diagnosis of cancer within past 5 years and/or currently undergoing treatment for any cancer.
* Any clinical condition, diagnosis, or social circumstance that, in the opinion of the Investigator, would be mean participation in the study would be contraindicated.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study will enroll sufficient subjects to yield a minimum of 60 subjects in Study Group 1, 30 subjects in Study Group 2 and 60 subjects in Study Group 3 - a total of 150 evaluable study subjects who meet all inclusion and exclusion criteria. Eligible subjects will be men and women age ≥ 18 years for Group 1 and 2 and 55 - 79 years inclusive for Group 3. Group 3 study subjects must also meet NLST guidelines of being at high risk for lung cancer: greater than or equal to a 30 pack year smoking history (equivalent of 1 pack per day for 30 or more years) and a current smoker or quit less than 15 years ago.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-08-13 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
The diagnostic performance of AminoIndex™ to discriminate lung cancer patients from high-risk subjects. | 6 months
  To evaluate the diagnostic performance characteristics of the AminoIndex™ technology among patients at high risk for developing lung cancer as compared with standard lung cancer screening and diagnostic procedures including low-dose CT, high-dose CT, biopsy and histopathology.

SECONDARY OUTCOMES:
The capability of AminoIndex™ to distinguish malignant lung cancer from benign lung nodules. | 6 months
Gathering residual patient samples that will be used for discovery research. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregg S. Britt, Study Director — Innovis LLC
Locations (3):
- United States (3):
  - Florida Lung Asthma and Sleep Specialists P.A., Celebration, Florida
  - Pulmonary and Critical Care Associates of Baltimore, Baltimore, Maryland
  - Vanderbilt-Ingram Cancer Center (VICC), Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No